CLINICAL TRIAL: NCT06052592
Title: Metabolomic Profile in Breastfed Late Preterm Infants Versus Standard Formula Milk or Postbiotic-supplemented Formula Milk
Brief Title: Metabolomic Profile in Breastfed Late Preterm Infants
Status: Completed | Type: Observational
Sponsor: Ospedale Buon Consiglio Fatebenefratelli (Other)
Collaborators: University of Salerno (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernardo, Head of Department of Woman and Child, Ospedale Buon Consiglio Fatebenefratelli
Other Study IDs: 1680/CE Lazio 1
Record Dates: First submitted 2023-08-03; First posted 2023-09-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-08

CONDITIONS: Formula Milk; Breast Milk Collection; Postbiotic Supplemented Formula Milk
Keywords: newborn; human milk; formula milk; postbiotic
MeSH Terms: conditions — Breast Milk Expression | interventions — Milk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: Newborns fed with formula milk supplemented with 20 mg/day of fermented FOS from Lactobacillus paracasei strain CNCM I-5220 and Vitamin D (0.5 ml of SMART D3 MATRIX)
  Interventions: Other: Milk
- Group B: Newborns fed with formula milk
  Interventions: Other: Milk
- Group C: Newborns fed with exclusive breast milk
  Interventions: Other: Milk

INTERVENTIONS:
Other: Milk — Newborns will be fed with breast milk, formula milk or postbiotic formula milk

SUMMARY:
Exclusive breast milk is recommended from birth to 6 months of life to promote the development of a balanced intestinal microbiota. Human milk provides several bioactive components, from natural probiotics such as Bifidobacterium spp. and Lactobacillus spp., to their metabolites which colonize the intestine of the newborn. However, if breast milk is not available or insufficient, it is used formula milk as a substitute. Infant formula can be supplemented with postbiotics to promote maturation of immune, metabolic and microbial components, similar to breast milk. Postbiotics are preparations composed of both microbial constituents and their metabolites, produced during fermentation.

DETAILED DESCRIPTION:
A balanced nutrition starting from early childhood significantly influences growth and psychomotor development. Exclusive breast milk is the recommended nutritional choice from birth to 6 months of life, as it guarantees everything necessary for growth, maturation, protection from infections, promoting the development of a balanced intestinal microbiota. Several prenatal and perinatal factors including the type of delivery, the use of antibiotics, diet and other environmental factors, can influence the microbial colonization of the newborn. Thus, it is generally accepted that the gut microbiota of the healthy, full-term, vaginally born, breastfed infant is the gold standard for a favorable microbial composition in the early years of life. Human milk provides several bioactive components, from natural probiotics such as Bifidobacterium spp. and Lactobacillus spp., to their metabolites ("natural postbiotics"), which colonize the intestine of the newborn. These metabolites regulate the development of the immune system and attenuate the inflammatory processes. However, if breast milk is not available or insufficient to meet the nutritional needs of the infant, formula milk is proposed and used as a substitute. Given the benefits, it is essential that infant formula is as close to human milk as possible, providing bioactive substances that target gut and immune system health. Current research focuses on optimizing artificial formulas, with the aim of resembling human milk in composition and functionality, with some on the market already including probiotics, prebiotics, synbiotics and postbiotics. However, it still remains to be clarified which is the best formulation and the exact consequences on the immune, metabolic and microbial system of the newborn. In particular, postbiotics are preparations composed of both microbial constituents and their metabolites, produced during fermentation. It has already been highlighted in the literature that the enrichment of formula milk with post-biotics would seem to offer advantages for feeding term infants. Furthermore, it promotes an immune, metabolic and microbial component maturation, similarly to human milk, thus making postbiotic supplements very promising and interesting in the nutrition of newborns and infants.

ELIGIBILITY:
Inclusion Criteria:

* Weight appropriate to gestational age (percentiles >10th and <90th)
* Written informed consent

Exclusion Criteria:

* Cardiological diseases
* Liver disease
* Gastrointestinal diseases with malabsorption
* Endocrinological diseases
* Perinatal infections
* Metabolic and genetic diseases
* Born to mothers with endocrinological and metabolic diseases
* Withdrawal of informed consent

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at Ospedale Buon Consiglio Fatebenefratelli, Naples
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of metabolomic profile by liquid chromatography mass spectrometry in breastfed late preterm infants | 5 days after delivery
  To detect the differences in the metabolome of the newborns
Evaluation of metabolomic profile by liquid chromatography mass spectrometry in breastfed late preterm infants | 1 month after delivery
  To detect the differences in the metabolome of the newborns
Evaluation of metabolomic profile by liquid chromatography mass spectrometry in breastfed late preterm infants | 3 months after delivery
  To detect the differences in the metabolome of the newborns

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, MD, Principal Investigator — Ospedale Buon Consiglio Fatebenefratelli
Locations (2):
- Italy (2):
  - Department of Pharmacy, University of Salerno, Salerno, Naples
  - Department of Woman and Child, Buon Consiglio Fatebenefratelli Hospital, Napoli, Napoli

IPD SHARING:
Plan to Share IPD: No